CLINICAL TRIAL: NCT05549687
Title: Randomized Control Trial of the Effect of an E-Health Support Program on Patient Reported Outcomes of Women Newly Diagnosed With Breast Cancer
Brief Title: E-Health Support Program (PACK Health Program) in Supporting Patient Reported Symptoms in Newly Diagnosed Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-0761; NCI-2019-02645 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0761 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2022-09-07; First posted 2022-09-22 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Pack Health Program) (Experimental): Patients participate in the Pack Health Program which includes up to 60 scheduled touch points via phone, text, email and a mobile application and weekly interaction with a health coach over 3 months. They also have access to standard of care support services at MD Anderson including a telephone triage line 5 days a week between 8 a.m. and 5 p.m.
  Interventions: Other: Questionnaire Administration; Procedure: Supportive Care
- Group II (standard of care support services) (Active Comparator): Patients receive standard of care support services with a telephone triage line available 5 days a week between 8 a.m. and 5 p.m.
  Interventions: Other: Questionnaire Administration; Procedure: Supportive Care

INTERVENTIONS:
Other: Questionnaire Administration — Ancillary studies
Procedure: Supportive Care — Participate in Pack Health, an electronic support program
  Arms: Group I (Pack Health Program)
Procedure: Supportive Care — Access to telephone triage line for support care services
  Other Names: Therapy, Supportive
  Arms: Group II (standard of care support services)

SUMMARY:
This trial studies how well an electronic (e)-health support program, called the PACK Health Program, supports patient reported symptoms in newly diagnosed patients with breast cancer. PACK Health offers a symptom management program involving both interpersonal interaction, as well as e-modules for patients diagnosed with cancer to better manage pain, fatigue, depression, anxiety, and to navigate care more effectively through e-health coaching and tools. Participating in the PACK Health Program may support breast cancer patients' reported side effects and experience of care during chemotherapy treatment and may ultimately improve overall health.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To examine the impact of an e-health support program on patient reported outcomes.

SECONDARY OBJECTIVES:

I. To evaluate the effect of e-health support program in comparison with standard of care support services, on the symptom experience of patients receiving chemotherapy in the ambulatory setting.

II. To evaluate the effect of e-health support program in comparison with standard of care support services, on the satisfaction of patients receiving chemotherapy in the ambulatory setting.

III. To evaluate the effect of e-health support program, in comparison with standard of care support services, on the frequency of emergency room visits and hospital admissions for patients receiving chemotherapy in the ambulatory setting.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients participate in the PACK Health Program which includes up to 60 scheduled touch points via phone, text, email and a mobile application, as well as weekly interaction with a health coach over 3 months. Patients also have access to standard of care support services at MD Anderson including a telephone triage line 5 days a week between 8 a.m. and 5 p.m.

GROUP II: Patients receive standard of care support services with a telephone triage line available 5 days a week between 8 a.m. and 5 p.m.

ELIGIBILITY:
Inclusion Criteria:

* English speaking.
* Newly diagnosed women with a breast cancer diagnosis preparing to undergo chemotherapy for the first time.
* All chemotherapy treatment to be completed at the study institution.
* Access to electronic resources, defined for the purposes of this study as a mobile phone, a landline phone, a computer, or another device with the capacity to receive calls, texts, or e-mails.

Exclusion Criteria:

* Patients who have received previous chemotherapy treatment for cancer.
* Patients who are unable to verbalize (e.g. due to tracheostomy).
* Patients enrolled on Protocol 2016-0300, as these patients will be receiving proactive triage calls from nurses that could skew their symptom reporting.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Impact of electronic (e)-health support program on patient reported outcomes | Baseline up to 3 months
  Measured with the National Institutes of Health Patient Reported Outcomes Measurement Information System (PROMIS) Global Health Scale. Summary statistics and box plots will be used to describe PROMIS scores by intervention arm and assessment time. A 2-sample t-test will be used to compare PROMIS scores at 3 months between intervention groups. Linear mixed effects models (LMMs) will be used to assess PROMIS scores over time. The models will include assessment time, intervention and baseline score as fixed effects and intercept as a random effect. Additional models will be created to include possible confounding covariates.
  PROMIS instrument scores will be reviewed and patients referred to the primary medical team if they score 1 on items 1-6, and 9, indicating poor health state and 4 or greater on items 8 and 10, indicating potential emotional distress or moderate to severe fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Hacker, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org